CLINICAL TRIAL: NCT02814747
Title: Preferences and Representations Concerning High-throughput Sequencing Technologies in Medical Genetics. The Case of Development Anomalies.
Brief Title: Evaluate and Understand Preferences and Representations in Families of Patients With Regard to High-throughput Sequencing Technology for Diagnostic Purposes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None
Other Study IDs: OLIVIER-FAIVRE 2014
Record Dates: First submitted 2016-06-16; First posted 2016-06-28 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Rare Diseases
MeSH Terms: conditions — Rare Diseases | interventions — Saline Solution, Hypertonic

ARMS (2):
- quantitive study: 500 patients likely to be candidates for HTS (Experimental): quantitive study: 500 patients likely to be candidates for HTS at CR in Dijon and Lyon, that is to say patients with development anomalies and/or intellectual deficiency with no etiological diagnosis.
  Interventions: Other: quantitive study: 500 patients likely to be candidates for HTS
- qualitative study: 30 patients who have benefited from HTS and (Experimental): qualitative study: 30 patients who have benefited from HTS and the medical geneticists who accompanied them in this approach.
  Interventions: Other: qualitative study: 30 patients who have benefited from HTS

INTERVENTIONS:
Other: quantitive study: 500 patients likely to be candidates for HTS
  Arms: quantitive study: 500 patients likely to be candidates for HTS
Other: qualitative study: 30 patients who have benefited from HTS
  Arms: qualitative study: 30 patients who have benefited from HTS and

SUMMARY:
After the use of DNA chips for diagnostic purposes, high-throughput sequencing (HTS) is transforming the field of developmental diseases, from fundamental research to care. Nonetheless, before HTS can be transferred to everyday clinical practice, in particular for expert diagnosis using exome HTS, it is necessary to anticipate the nature of the information to be given to patients and to parents in order to obtain consent for exome HTS.

The objective in terms of public health is to allow patients with rare diseases to benefit from innovative technologies in optimal conditions of information and accompaniment.

the objectives of this project are to

1. evaluate the preferences of families of patients with development disorders as regard to suspicious and incidental findings from HTS before its introduction for diagnostic purpose,
2. and then, following the exome analyses carried out for diagnostic purposes, describe, analyse and understand the experience, expectations and reactions of families and geneticists concerning the diagnostic trajectory in general and at the time the results of the HTS were announced in particular A methodology that associated quantitative and qualitative approaches was chosen so as to combine the advantages and overcome the shortcomings of each: a quantitative study to investigate a large number of patients, which would ensure a certain representativeness of the population and allow sub-groups analyses to study the upstream phase concerning indications for high-throughput sequencing; and a qualitative study, which though it allows only a small number of patients to be investigated, makes it possible to describe, analyze and understand in depth the complex downstream phenomena of high-throughput sequencing results

ELIGIBILITY:
Quantitative study

* INCLUSION CRITERIA

  * parents of patients with development anomaly and/or intellectual deficiency with no etiological diagnosis
  * parents of patients consulting at the centres of reference in Dijon or Lyon
  * parents of patients who have not already benefited from HTS
  * parents of patients who are fluent in French
* NON-INCLUSION CRITERIA

  * persons without national health insurance cover
  * inability to answer the questionnaires

Qualitative study

* INCLUSION CRITERIA

  * persons who have provided written informed consent
  * parents of patients with a development anomaly
  * parents of patients consulting at the centres of reference in Dijon or Lyon
  * parents of patients who have already benefited from HTS for diagnostic purposes
  * persons fluent in French
* NON-INCLUSION CRITERIA

  * persons without national health insurance cover
  * cognitive impairment making it impossible for the person to understand the aims of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Preferences of families of patients concerning the diffusion of incidental results with uncertain interpretation from high-throughput sequencing prior to whole exome analyses | day one

SECONDARY OUTCOMES:
Questionnaire on the experiences, expectations and reactions of families and geneticists with regard to the moment the results are announced | day one

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Chassagne A, Pelissier A, Houdayer F, Cretin E, Gautier E, Salvi D, Kidri S, Godard A, Thauvin-Robinet C, Masurel A, Lehalle D, Jean-Marcais N, Thevenon J, Lesca G, Putoux A, Cordier MP, Dupuis-Girod S, Till M, Duffourd Y, Riviere JB, Joly L, Juif C, Putois O, Ancet P, Lapointe AS, Morin P, Edery P, Rossi M, Sanlaville D, Bejean S, Peyron C, Faivre L. Exome sequencing in clinical settings: preferences and experiences of parents of children with rare diseases (SEQUAPRE study). Eur J Hum Genet. 2019 May;27(5):701-710. doi: 10.1038/s41431-018-0332-y. Epub 2019 Feb 1. PMID 30710147